CLINICAL TRIAL: NCT03075033
Title: The Shikani Optical Stylet As An Alternative To Awake Fiberoptic Intubation In Patients At Risk Of Secondary Cervical Spine Injury - A Randomized Controlled Trial.
Brief Title: SOS Versus Awake Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Rabab Sber Saleh Mahrous, principal investigator, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shikani2017
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Cervical Spine Instability
Keywords: Shikani optical stylet, rigid optical stylets, awake, fiber-optic intubation, and cervical spine injury.

STUDY DESIGN:
Intervention Model Description: This prospective, randomized study was approved by the local ethical committee of Alexandria main university hospital. Written informed consent was obtained from all the participants. Sixty patients aged 18-65 year with American Society of Anaesthesiologists physical status I-III with a neurosurgical diagnosis of cervical instability or at risk of secondary cervical injury, who were scheduled for awake intubation and self-positioning prone for elective neurological intervention, were enrolled in this study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOS gruop (Active Comparator): Use of The Shikani Optical Stylet In Patients At Risk Of Secondary Cervical Spine Injury
  Interventions: Device: Shikani optical stylet
- Awake Fiberoptic Intubation (Active Comparator): Use of Awake Fiberoptic Intubation In Patients At Risk Of Secondary Cervical Spine Injury
  Interventions: Device: Flexible fiberoptic bronchoscope for

INTERVENTIONS:
Device: Shikani optical stylet — Tracheal intubation is performed using Shikani optical stylet. The shikani optical stylet was bent to the same bend as a Mackintosh laryngoscope blade, lubricated and the endotracheal tube was mounted on it. The tube was settled to the stylet by the 'adjustable tube stop' so that the tip of the stylet did not project beyond the end of the tube. After intubation the 'tube stop' was released and the tube was unmounted into the trachea; the stylet was removed.
  Arms: SOS gruop
Device: Flexible fiberoptic bronchoscope for — AwakeRracheal intubation using flexible fiberoptic bronchoscope in patients with cervical spine instability
  Arms: Awake Fiberoptic Intubation

SUMMARY:
Background: Conventional intubation of the trachea and consequent prone positioning of anaesthetized patients with cervical spine instability may result in secondary neurological injury. Historically, the flexible fiber-optics used to be the chief choice for patients presenting with cervical spine instability surgery either with normal, predicted difficult airway, or even unanticipated difficult airway. Recently, the rigid optical stylets have shown promise in assisting difficult intubations.

Purpose: The aim of the present study was to compare the efficacy of Shikani optical stylet (SOS) with the flexible fiberscope for awake intubation in patients with cervical spine instability.

Methods: Sixty adult patients with a neurosurgical diagnosis of cervical instability or at risk of secondary cervical injury, who were planned for awake intubation and self-positioning prone, were registered in this study and were randomly categorized into two equal groups (thirty patients each), a fiberoptic group and a SOS group, then assessment of coughing and gagging during and after intubation, time to intubation, number of attempts for successful intubation, haemodynamic parameters, careful examination of the oropharynx to determine any lip or mucosal trauma, and eventually the motor function by the ability to move arms and legs were assessed after tracheal intubation and after positioning prone.

DETAILED DESCRIPTION:
Aim of the work:

The aim of this study was to compare the efficacy of shikani optical stylet with the flexible fiberoptic bronchoscope for awake intubation in patients with cervical spine instability.

Patients and Methods:

This prospective, randomized study was approved by the local ethical committee of Alexandria main university hospital. Written informed consent was obtained from all the participants. Sixty patients aged 18-65 year with American Society of Anaesthesiologists physical status I-III with a neurosurgical diagnosis of cervical instability or at risk of secondary cervical injury, who were scheduled for awake intubation and self-positioning prone for elective neurological intervention, were enrolled in this study. Patients with increased risk of pulmonary aspiration, requirement for rapid sequence induction or associated head injury precluding adequate clinical neurological examination were excluded from the study. All patients received rigid neck collar. Data collected from each patient included demographic data, level of cervical spine pathology and the neurological status.

An assistant who wasn't concerned within this study got numbered opaque pre-sealed envelopes containing the randomised group allocations after every patient was joined into the study. Patients were randomly assigned into either a fiberoptic group (30) or a Shikani group (30) utilizing a sealed-envelope technique.

Anaesthetists concerned within the study had expertise with both devices and were assured in consuming the devices in a difficult airway situation.

Routin pre-anaesthetic assessments were performed, in addition to a standard airway assessment, recording the presence of any oro-pharyngeal injury before surgery. Non-invasive monitoring was used before intubation comprising pulse oximetry, blood pressure and electrocardiography. Before starting topical anaesthesia, all patients were given atropine 0.4 mg as an anti sialagogue agent, midazolam 2 mg and increments of fentanyl 25mic intravenously till the patient is calm and sedated but controlling his airway.

Topical anaesthesia of the oral cavity was performed with lidocaine 10% spray. Anesthesia of the larynx just above the vocal cords, vocal cords and the upper trachea was encountered with superior laryngeal nerves block using 4 ml of 2% lidocaine (2 ml on each side), at the lateral ends of the thyrohyoid membrane just beneath the greater cornu of the hyoid bone and recurrent laryngeal nerve block (Trans-tracheal injection) using a 20-gauge plastic catheter, 4ml of 2% lidocaine through the cricothyroid membrane at the end of inspiration.

Tracheal intubation was then executed with either the flexible fiberoptic bronchoscope or the Shikani optical stylet, according to the randomised allocation. The shikani optical stylet was bent to the same bend as a Mackintosh laryngoscope blade, lubricated and the endotracheal tube was mounted on it. The tube was settled to the stylet by the 'adjustable tube stop' so that the tip of the stylet did not project beyond the end of the tube. The anaesthetist hold and elevated the mandible using the left hand, the patient was asked to protrude his tongue if applicable and the stylet was introduced into the right side of the mouth and advanced until the tip was in hypopharynx. Then, under direct vision the tip was inserted between the vocal cords.The 'tube stop' was released and the tube was unmounted into the trachea; the stylet was removed. Once tracheal intubation was accomplished, confirmation of the position of endotracheal tube by capnography and chest auscultation. The patients were then asked to move to the prone position on the bolsters, in the cases planned for posterior approach of the cervical spine. The anaesthesia provider guarded the head and tube during the move and neurological examination was repeated. Once the position is settled, the presence of end tidal carbon dioxide was confirmed and general anaesthesia was set up.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists physical status I-III with a neurosurgical diagnosis of cervical instability or at risk of secondary cervical injury, who were scheduled for awake intubation and self-positioning prone for elective neurological intervention

Exclusion Criteria:

* Patients with increased risk of pulmonary aspiration, requirement for rapid sequence induction or associated head injury precluding adequate clinical neurological examination were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Coughing and gagging | during and after intubation
  using a scale of 1 to 4: (1= none; 2 < 3 times (slight coughing and gagging comparable to "clearing ones throat"); 3 > 2 times (mild coughing or gagging lasting less than a minute); 4 = persistent coughing or gagging]
Time to intubation | the interval from the start of intubation to the completion of intubation
  Measure the time in minutes from the start of intubation to the completion of intubation
Number of attempts for successful intubation | During intubation
  How many trials were taken till achieve the intubation
The changes in the haemodynamic parameters | Pre-induction, pre-intubation and at 3 and 5 min after intubation
  the haemodynamic parameters including: heart rate, systolic and diastolic blood pressures during the intubation process with readings taken pre-induction, pre-intubation and at 3 and 5 min after intubation.

IPD SHARING:
Plan to Share IPD: No